CLINICAL TRIAL: NCT00908596
Title: Prospective Non-randomized (Pharmacoepidemiologic) Cohort Study (Open-label, Multicenter) to Assess the Magnitude of Potential Risk With the Administration of Primovist/Eovist in Patients With Moderate to Severe Renal Impairment for the Development of Nephrogenic Systemic Fibrosis (NSF) Based on Diagnostically Specific Clinical and Histopathologic Information.
Brief Title: Primovist / Eovist in Renally Impaired Patients
Acronym: PERI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13701; 2008-005867-33 (EudraCT Number)
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Contrast Media
Keywords: Nephrogenic Systemic Fibrosis (NSF); Primovist / Eovist
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadoxetic acid disodium (Primovist/Eovist, BAY86-4873) (Experimental): Participants received Primovist at a dose of 0.025 mmol/kg body weight (BW) intravenously.
  Interventions: Drug: Gadoxetic acid disodium (Primovist, BAY86-4873)

INTERVENTIONS:
Drug: Gadoxetic acid disodium (Primovist, BAY86-4873) — Primovist/Eovist in approved indications at approved dosages

SUMMARY:
Patients with moderate to severe renal impairment scheduled for a magnetic resonance imaging (MRI) scan and injection with a contrast agent, Primovist/Eovist, will be asked to participate.

The administration of contrast agents that contain gadolinium such as Primovist/Eovist might increase a potential risk to develop a rare condition called nephrogenic systemic fibrosis (NSF) in patients with renal impairment. This study is to assess the potential risk to develop NSF in patients with renal impairment after the administration of Primovist/Eovist.

Patients who are enrolled in this study will receive a Primovist/Eovist enhanced MRI scan which was prescribed by the referring doctor. After the MRI scan the patient will be included in a two year follow-up period to assess if signs or symptoms suggestive of NSF have appeared.

DETAILED DESCRIPTION:
Adverse events data will be reported in Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be scheduled for Contrast enhanced magnetic resonance imaging (CE-MRI) of the liver with Primovist/Eovist based on careful risk/benefit evaluation at the recommended dose in one of the approved indications
* Patient must fulfill criteria for moderate (Estimated glomerular filtration rate [eGFR] 30 - 59 mL/min/1.73 m^2) to severe (eGFR < 30 mL/min/1.73 m^2) renal impairment.

Exclusion Criteria:

* Gadolinium based contrast agent (GBCA)-enhanced MRI (or administration of a GBCA for any other CE imaging procedure) other than Primovist/Eovist within 12 months prior to administration of Primovist/Eovist
* History of existing NSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2009-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (46):
- United States (12):
  - Los Angeles, California
  - Jacksonville, Florida
  - Honolulu, Hawaii
  - Topeka, Kansas
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Brooklyn, New York
  - New York, New York
  - Durham, North Carolina
  - Memphis, Tennessee
  - Houston, Texas
  - San Antonio, Texas
- Australia (5):
  - Herston, Queensland
  - Woollongabba, Queensland
  - Adelaide, South Australia
  - Geelong, Victoria
  - Westmead NSW
- Austria (2):
  - Graz
  - Vienna
- Germany (12):
  - Heidelberg, Baden-Wurttemberg
  - Stuttgart, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Hanover, Lower Saxony
  - Dortmund, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Dresden, Saxony
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Gera, Thuringia
- Italy (8):
  - Rozzano, Milano
  - Pozzuoli, Napoli
  - Candiolo, Torino
  - Brescia
  - Milan
  - Napoli
  - Palermo
  - Pisa
- South Korea (3):
  - Busan, South Korea
  - Seoul, South Korea
  - Seoul
- Granada, Granada, Spain
- Thailand (2):
  - Bangkok
  - Songkhla
- Bristol, United Kingdom

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant's first visit was on 21 May 2009. 35 study centers in Australia, Austria, Germany, Italy, Spain, South Korea, UK, USA, and Thailand screened and enrolled participants scheduled to undergo contrast enhanced magnetic resonance imaging (CE-MRI) of the liver with Primovist/Eovist within the approved indications.
Pre-assignment Details: A total of 364 participants were enrolled. Of these, 4 were withdrawn prior to magnetic resonance imaging (MRI) already since they failed to meet the study entrance criteria, and 3 were withdrawn for other reasons. Participants had to have moderate to severe renal impairment (estimated glomerular filtration rate [eGFR] 65 mL/min/1.73 m^2 or less).
Groups:
- Gadoxetic Acid Disodium - Mild Renal Impairment: Participants with eGFR (estimated glomerular filtration rate) prior to Primovist/Eovist injection >65 mL/min/1.73 m^2. Participants received Primovist/Eovist as part of their routine medical care.
- Gadoxetic Acid Disodium - Extended Moderate Renal Impairment: Participants with eGFR prior to Primovist/Eovist injection between > 59 and ≤ 65 mL/min/1.73 m^2. Participants received Primovist/Eovist as part of their routine medical care.
- Gadoxetic Acid Disodium - Moderate Renal Impairment: Participants with eGFR prior to Primovist/Eovist injection between ≥ 30 and ≤ 59 mL/min/1.73 m^2. Participants received Primovist/Eovist as part of their routine medical care.
- Gadoxetic Acid Disodium - Severe Renal Impairment: Participants on dialysis or if not on dialysis with eGFR prior to Primovist/Eovist injection < 30 mL/min/1.73 m^2. Participants received Primovist/Eovist as part of their routine medical care.
Period: Overall Study
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Started | 47 | 32 | 193 | 85
Completed | 0 | 19 | 119 | 48
Not Completed | 47 | 13 | 74 | 37
Not completed — Other reasons | 46 | 6 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 12 | 4
Not completed — Death | 0 | 5 | 57 | 32
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment | Total
Number analyzed (Participants) | 47 | 32 | 193 | 85 | 357
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (9.55) | 65.3 (12.03) | 65.5 (10.88) | 62.2 (13.83) | 64.7 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 7 | 46 | 30 | 103
  Male | 27 | 25 | 147 | 55 | 254
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 15 | 9 | 101 | 63 | 188
  Black | 2 | 1 | 6 | 2 | 11
  Hispanic | 0 | 1 | 3 | 0 | 4
  Asian | 27 | 16 | 56 | 8 | 107
  other | 3 | 5 | 27 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate to Severe Renal Impairment, Who Develop NSF (Nephrogenic Systemic Fibrosis), Based on Diagnostically Specific Clinical and Histopathological Information
Description: A diagnosis of NSF was assumed for subjects with a minimum combined clinical (scale: 0-other diagnosis, 1-inconsistent, 2-suggestive, 3-consistent, 4-highly consistent) and histopathological score (same scale as clinical score). Either the clinical score or the histopathology score had to be at least 2, and the other at least 3.
Time Frame: Up to 24 months following the administration of Primovist/Eovist
Population: Full Analysis Set: all participants who were enrolled and received Primovist/Eovist
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Number analyzed (Participants) | 47 | 32 | 193 | 85
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Moderate to Severe Renal Impairment in Whom no Biopsy Was Obtained Who Develop NSF-like Symptoms Based on Diagnostically Specific Clinical Information Summarized by Clinical Score
Description: Participants in whom no biopsy was obtained with a clinical score of 4 on a scale comprising 0-other diagnosis, 1-inconsistent, 2-suggestive, 3-consistent, 4-highly consistent.
Time Frame: Up to 24 months following the administration of Primovist/Eovist
Population: Full Analysis Set: all participants who were enrolled and received Primovist/Eovist
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Number analyzed (Participants) | 47 | 32 | 193 | 85
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Confidence of the Investigator to Make a Diagnosis Based on the Primovist/Eovist Enhanced MRI (Magnetic Resonance Imaging)
Description: The investigator was to record his / her confidence in making a diagnosis using a 4 point scale (Very high confidence / High confidence / Moderate / Low confidence). For some participants the values were not collected.
Time Frame: Immediately after Primovist/Eovist-enhanced MRI
Population: Full Analysis Set: all participants who were enrolled and received Primovist/Eovist
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Number analyzed (Participants) | 47 | 32 | 193 | 85
Participants
  Very high | 26 | 16 | 98 | 33
  High | 15 | 13 | 80 | 38
  Moderate | 5 | 3 | 12 | 4
  Low | 1 | 0 | 2 | 1

4. Secondary Outcome: Number of Participants With "Excellent / Good / Adequate / Insufficient" Scores for Lesion Detection
Description: The investigator was to record the imaging efficacy by evaluation of lesion detection using a 4 point scale (Excellent / Good / Adequate / Insufficient). For some participants the values were not collected.
Time Frame: Immediately after Primovist/Eovist-enhanced MRI
Population: Full Analysis Set: all participants who were enrolled and received Primovist/Eovist
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Number analyzed (Participants) | 47 | 32 | 193 | 85
Participants
  Excellent | 29 | 20 | 99 | 34
  Good | 15 | 12 | 74 | 29
  Adequate | 1 | 0 | 15 | 8
  Insufficient | 0 | 0 | 1 | 2

5. Secondary Outcome: Number of Participants With "Excellent / Good / Adequate / Insufficient" Scores for Lesion Delineation
Description: The investigator was to record the imaging efficacy by evaluation of lesion delineation using a 4 point scale (Excellent / Good / Adequate / Insufficient). For some participants the values were not collected.
Time Frame: Immediately after Primovist/Eovist-enhanced MRI
Population: Full Analysis Set: all participants who were enrolled and received Primovist/Eovist
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Number analyzed (Participants) | 47 | 32 | 193 | 85
Participants
  Excellent | 27 | 16 | 94 | 31
  Good | 15 | 16 | 77 | 34
  Adequate | 3 | 0 | 16 | 6
  Insufficient | 0 | 0 | 1 | 3

6. Secondary Outcome: Number of Participants With "Excellent / Good / Adequate / Insufficient" Scores for Lesion Characterization
Description: The investigator was to record the imaging efficacy by evaluation of lesion characterization using a 4 point scale (Excellent / Good / Adequate / Insufficient). For some participants the values were not collected.
Time Frame: Immediately after Primovist/Eovist-enhanced MRI
Population: Full Analysis Set: all participants who were enrolled and received Primovist/Eovist
Measure: Number; unit: Participants
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Number analyzed (Participants) | 47 | 32 | 193 | 85
Participants
  Excellent | 30 | 13 | 93 | 33
  Good | 12 | 16 | 79 | 34
  Adequate | 2 | 3 | 14 | 5
  Insufficient | 1 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to 24 months following the administration of Primovist/Eovist
Arm/Group | Gadoxetic Acid Disodium - Mild Renal Impairment | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment | Gadoxetic Acid Disodium - Moderate Renal Impairment | Gadoxetic Acid Disodium - Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/32 | 0/193 | 1/85
Other Adverse Events (participants affected / at risk) | 0/47 | 1/32 | 7/193 | 6/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadoxetic Acid Disodium - Mild Renal Impairment (N=47) | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment (N=32) | Gadoxetic Acid Disodium - Moderate Renal Impairment (N=193) | Gadoxetic Acid Disodium - Severe Renal Impairment (N=85)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gadoxetic Acid Disodium - Mild Renal Impairment (N=47) | Gadoxetic Acid Disodium - Extended Moderate Renal Impairment (N=32) | Gadoxetic Acid Disodium - Moderate Renal Impairment (N=193) | Gadoxetic Acid Disodium - Severe Renal Impairment (N=85)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 1
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was stopped early since the FDA released the sponsor from completing enrollment because the NSF incidence estimate was lower than the original literature-based estimate, and since enrollment quota were not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less